CLINICAL TRIAL: NCT02938195
Title: Phase II Study of Optimum Design of Neo-adjuvant Chemoradiotherapy Followed by Surgery for Squamous Cell Esophageal Cancer
Brief Title: Phase II Study of Neo-adjuvant Chemoradiotherapy for Squamous Cell Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate chief physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHEC001
Record Dates: First submitted 2016-10-15; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Cancer; Chemoradiation; Surgery
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental arm (Experimental): PF regimen (cis-platinum of 25 mg/m2/d, d1-3; 5-fluorouracil of 500mg/m2/d, d1-4) every 4 weeks for 2 cycles concurrently with three-dimensional radiation therapy or intensity-modulated radiotherapy followed by surgery 4-8weeks after neoadjuvant therapy in a standard manner.
  Interventions: Radiation: radiotherapy; Procedure: Surgery

INTERVENTIONS:
Radiation: radiotherapy — The clinical target volume of radiotherapy only includes the visible tumor and lymph nodes and the investigators wouldn't do any prophylactic radiation treatment.
Procedure: Surgery — Surgery would be done 4-8 weeks after neoadjuvant chemoradiotherapy.

SUMMARY:
The investigators designed a new preoperative chemoradiotherapy regimen to focus on the most important radiation area and hope to reduce the radiation volume and try to reduce the postoperative mortality and treatment-related mortality.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is the eighth most common cancers in the world, with more than 480,000 new cases and 400,000 deaths occurred annually worldwide. In China, either new cases or deaths account for more than half of the world. Morever, over 90% of Chinese patients have esophageal squamous cell carcinoma (ESCC).

Surgery is the main treatment of this disease, but the prognosis of patients with locally advanced esophageal cancer is rather poor. As a result of surgery alone, the 5-year survival rate of about 25% has not changed significantly in several decades.

Neo-adjuvant chemoradiotherapy followed by surgery seems hopeful to improve the survival of EC. Recently, the CROSS trial has demonstrated that preoperative chemoradiotherapy can significantly increased the overall survival of patients with EC compared with surgery alone. However,a recent meta-analysis has indicated that an increased risk of postoperative mortality and treatment-related mortality was apparent in ESCC with the treatment of neo-adjuvant chemoradiotherapy.

Compare to surgery alone,the advantage of neoadjuvant chemoradiotherapy is reflected in the significantly higher percentage of R0 resections and higher rate of pathological complete response.

Thus,the investigators designed a new preoperative chemoradiotherapy regimen to focus on the most important radiation area and hope to reduce the radiation volume and try to reduce the postoperative mortality and treatment-related mortality.

Radiotherapy:Patients will be conducted CT simulation, and three-dimensional radiation therapy or Intensity-modulated radiation therapy was performed. 1.8Gy/fraction, 5 fractions a week, with a total dose of 4140cgy will be delivered for all patients by 6-MV-X-ray of linear accelerator.

Chemotherapy:Patients will be concurrently administered with irradiation every 4 weeks with PF regimen (cis-platinum of 25 mg/m2/d, d1-3; 5-fluorouracil of 500mg/m2/d, d1-4) for 2 cycles.

Surgery:Patients will receive operation 4-8 weeks after chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of squamous cell thoracic esophageal carcinoma of Stage IIB or III, which is potentially resectable.
2. Patients must not have received any prior anticancer therapy.
3. More than 6 months of expected survival.
4. Age ranges from 18 to 70 years.
5. Absolute white blood cells count ≥4.0×109/L, neutrophil ≥1.5×109/L, platelets ≥100.0×109/L, hemoglobin ≥90g/L, and normal functions of liver and kidney.
6. Karnofsky performance status (KPS) of 90 or more.
7. Signed informed consent document on file.

Exclusion Criteria:

1. Patients are diagnosed or suspected to be allergic to cisplatin or 5-Fu.
2. Patients with concomitant hemorrhagic disease.
3. Pregnant or breast feeding.
4. Inability to use gastric conduit after esophagectomy because of a prior surgery.
5. Patients with concomitant peripheral neuropathy, whose CTC status is 2 or even more.
6. Have a prior malignancy other than esophageal carcinoma, carcinoma in situ of the cervix, nonmelanoma skin cancer or cured early stage of prostate cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients completing adjuvant chemoradiotherapy and surgery | 4-8weeks after surgery

SECONDARY OUTCOMES:
Percentage of R0 resection | 4-8weeks after surgery
Percentage of pathological complete response | 4-8weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Fu, Ph.D, Study Director — Department of Radiation Oncology,Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Background] Huang TC, Hsu CH, Lin CC, Tu YK. Systematic review and network meta-analysis: neoadjuvant chemoradiotherapy for locoregional esophageal cancer. Jpn J Clin Oncol. 2015 Nov;45(11):1023-8. doi: 10.1093/jjco/hyv119. Epub 2015 Aug 5. PMID 26246479
- [Background] Martinek J, Akiyama JI, Vackova Z, Furnari M, Savarino E, Weijs TJ, Valitova E, van der Horst S, Ruurda JP, Goense L, Triadafilopoulos G. Current treatment options for esophageal diseases. Ann N Y Acad Sci. 2016 Oct;1381(1):139-151. doi: 10.1111/nyas.13146. Epub 2016 Jul 8. PMID 27391867
- [Background] Ikebe M, Morita M, Yamamoto M, Toh Y. Neoadjuvant therapy for advanced esophageal cancer: the impact on surgical management. Gen Thorac Cardiovasc Surg. 2016 Jul;64(7):386-94. doi: 10.1007/s11748-016-0655-y. Epub 2016 May 10. PMID 27165288
- [Background] Purwar P, Bambarkar S, Jiwnani S, Karimundackal G, Laskar SG, Pramesh CS. Multimodality management of esophageal cancer. Indian J Surg. 2014 Dec;76(6):494-503. doi: 10.1007/s12262-014-1163-x. Epub 2014 Sep 11. PMID 25614726
- [Background] Kumagai K, Rouvelas I, Tsai JA, Mariosa D, Klevebro F, Lindblad M, Ye W, Lundell L, Nilsson M. Meta-analysis of postoperative morbidity and perioperative mortality in patients receiving neoadjuvant chemotherapy or chemoradiotherapy for resectable oesophageal and gastro-oesophageal junctional cancers. Br J Surg. 2014 Mar;101(4):321-38. doi: 10.1002/bjs.9418. Epub 2014 Feb 3. PMID 24493117